CLINICAL TRIAL: NCT00178113
Title: Phase I Clinical Trial: Randomized Lycopene Supplementation in Tobago Men With High-Grade Prostatic-Intraepithelial Neoplasia
Brief Title: A Pilot Study of Lycopene Supplementation in Prostatic Intraepithelial Neoplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA084950-05S1 (NIH); P200202-134PRC02-134
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Prostatic Intraepithelial Neoplasia
Keywords: Prostatic Intraepithelial Neoplasia; Prostate-Specific Antigen; lycopene
MeSH Terms: conditions — Prostatic Intraepithelial Neoplasia | interventions — Lycopene; Dietary Supplements; Geritol; Minerals

INTERVENTIONS:
Drug: - Lyc-O-Mato (dietary supplement, 30 mg lycopene/day)
Drug: - Certagen (multivitamins with minerals)

SUMMARY:
The purpose of this study is to determine whether dietary lycopene supplementation lowers serum prostate specific antigen(PSA) in men with high grade intraepithelial neoplasia (HGPIN).

DETAILED DESCRIPTION:
Observational studies suggest higher lycopene intake or higher lycopene blood levels are associated with a lower risk for prostate cancer. Two recent trials of lycopene supplementation conducted in men with prostate cancer, during the three weeks prior to radical prostatectomy, found a reduction in serum PSA suggesting a regression of prostate cancer.

High grade intraepithelial neoplasia (HGPIN)is thought to be a precancerous lesion, and men with HGPIN have an elevated risk of prostate cancer diagnosis on subsequent biopsy. The objective of this study is to determine whether dietary lycopene supplementation lowers serum prostate specific antigen(PSA)over four months of supplementation. Serum PSA is compared in men randomized to 30 mg/day lycopene plus a standard multivitamin versus standard multivitamin alone.

ELIGIBILITY:
Inclusion Criteria:

* biopsy reported high grade prostatic intraepithelial neoplasia
* and/or biopsy reported atypia
* and/or persistently elevated serum prostate specific antigen with normal biopsy

Exclusion Criteria:

* biopsy diagnosed prostate cancer
* serum prostate specific antigen > 40 ng/ml
* hospitalization in past six months
* history of allergy to tomatoes
* history of allergic dermatitis
* serious concurrent illness
* inability to provide informed consent

Ages: 40 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-07; Study Completion 2004-07

PRIMARY OUTCOMES:
Serum PSA at randomization, one month, four months

SECONDARY OUTCOMES:
Serum lycopene at randomization, one month, four months

CONTACTS AND LOCATIONS:
Overall Officials: Clareann H Bunker, PhD, Principal Investigator — University of Pittsburgh; Lewis H Kuller, MD, Study Director — University of Pittsburgh
Locations (1):
- Tobago Prostate Survey Office, Scarborough, Tobago, Trinidad and Tobago